CLINICAL TRIAL: NCT07005453
Title: Diagnostic Performance and Sustainability of Using SCALE-EYE During Real-Time Colonoscopy
Brief Title: Accuracy and Sustainability of SCALE-EYE Evaluation for Measuring Reliable Polyp Size
Acronym: ASSEMBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Peter Siersema, Prof. Dr. P.D. Siersema, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MEC-2024-0789
Record Dates: First submitted 2025-05-01; First posted 2025-06-05 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Polyps
Keywords: virtual scale endoscopy; biopsy forceps; optical assessment; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be split in two groups who will in parallel to each other undergo both SCALE-EYE measurement and biopsy-forceps assisted measurement, but there will be randomization in the order of measuring. So approximately half of the participants, in whom polyps are found, will first undergo SCALE-EYE measurement and then biopsy-forceps assisted measurement, and the other half of the participants will first undergo biopsy-forceps assisted measurement and then SCALE-EYE measurement.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCALE-EYE measurement than biopsy-forceps assisted measurement (Other): When colorectal polyps are identified, then first the polyp size is categorized by optical assessment by the endoscopist. Then the polyp size is categorized by SCALE-EYE measurement and afterwards by biopsy-forceps assisted measurement.
  Interventions: Device: SCALE-EYE (1)
- Biopsy-forceps assisted measurement than SCALE-EYE measurement (Other): When colorectal polyps are identified, then first the polyp size is categorized by optical assessment by the endoscopist. Then the polyp size is categorized by biopsy-forceps assisted measurement and afterwards by SCALE-EYE measurement.
  Interventions: Device: SCALE-EYE (2)

INTERVENTIONS:
Device: SCALE-EYE (1) — Participants will undergo the colonoscopy and once a colorectal polyp is identified, the polyp will first be measured by optical assessment by the endoscopist, then with SCALE-EYE and lastly by biopsy-forceps assisted measurement.
  Arms: SCALE-EYE measurement than biopsy-forceps assisted measurement
Device: SCALE-EYE (2) — Participants will undergo the colonoscopy and once a colorectal polyp is identified, the polyp will first be measured by optical assessment by the endoscopist, then by biopsy-forceps assisted measurement and lastly with SCALE-EYE.
  Arms: Biopsy-forceps assisted measurement than SCALE-EYE measurement

SUMMARY:
A multicenter, randomized, parallel group, endoscopist blinded study to assess the diagnostic performance and sustainability of SCALE-EYE in a screening and surveillance colonoscopy population.

Sustainability will be evaluated in terms of the reduction in colonoscopies, associated waste and carbon footprint.

DETAILED DESCRIPTION:
Objective: This study aims to assess the diagnostic performance of SCALE-EYE in a screening and surveillance colonoscopy population. Also, sustainability of SCALE-EYE in terms of the reduction in colonoscopies, associated waste and carbon footprint is evaluated.

Study design: A multicenter, randomized, parallel group, endoscopist blinded study.

Study population: The unit of analysis is the colorectal polyp rather than the participants, approximately 289 colorectal polyps are planned to be included. Based on an expected detection rate of roughly 1.20 polyps per colonoscopy in the study population, approximately 241 participants aged 55-80 years old, who are referred for screening or surveillance colonoscopy at the participating study sites and have signed the informed consent form (ICF), will be included into the study. Polyps of all shapes (flat, sessile, pedunculated) that are found during colonoscopy and are smaller than 25 mm, as judged by the endoscopist using optical assessment, are considered eligible for inclusion.

Intervention: Participants will undergo the colonoscopy and once a colorectal polyp is identified, the polyp will first be measured by optical assessment by the endoscopist and then in a randomized order measured by biopsy-forceps assisted measurement and SCALE-EYE measurement.

Primary outcome measurement: The diagnostic performance of SCALE-EYE for polyp size categorization during real-time colonoscopy in comparison to polyp size categorization with biopsy-forceps assisted measurement (the reference standard). This will be measured by accuracy, sensitivity, and specificity of SCALE-EYE categorization compared to size measurement with the reference standard.

Secondary outcome measurements:

* The diagnostic performance of SCALE-EYE for polyp size categorization during real-time colonoscopy in comparison to optical assessment by endoscopists for polyp size measurement.
* Sustainability (reduction of colonoscopies, the colonoscopy-associated waste and carbon footprint).
* The learning curve, this will be evaluated by exploring the association between the number of measurements performed and the time needed for measurement and experienced difficulty.
* The level of agreement between the endoscopist advised surveillance interval as based on SCALE-EYE, optical assessment, and the reference standard.
* Safety, in terms of (serious) adverse events up to 30 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 55-80
* Scheduled for fecal immunochemical test (FIT) screening or surveillance colonoscopy
* Polyps of all forms ≤25 mm as assessed by the endoscopist

Exclusion Criteria:

* No detected colorectal polyps or only diminutive (≤5 mm) hyperplastic rectal polyps are present
* Inadequate bowel preparation (Boston Bowel Preparation Score (BBPS) <2 per segment)
* Intraprocedural complications, not caused by the study device
* Known or suspected inflammatory bowel disease (IBD)
* Polyposis syndromes (e.g. serrated polyposis, familial adenomatous polyposis)
* Ileoanal pouch and anastomosis
* History of radiation or chemotherapy for colorectal lesions
* Scheduled for therapeutic procedure (for example intervention to stop a lower gastro-intestinal bleeding, endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD))
* Pregnancy
* No Informed consent (IC) possible

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
SCALE-EYE diagnostic performance versus biopsy-forceps | Immediately after the screening and/or surveillance colonoscopy
  The diagnostic performance of SCALE-EYE for polyp size categorization during real-time colonoscopy in comparison to polyp size categorization with biopsy-forceps assisted measurement (the reference standard). This will be measured by accuracy, sensitivity, and specificity of SCALE-EYE categorization compared to size measurement with the reference standard.

SECONDARY OUTCOMES:
SCALE-EYE diagnostic performance versus optical assessment | Immediately after the screening and/or surveillance colonoscopy
  The diagnostic performance of SCALE-EYE for polyp size categorization during real-time colonoscopy in comparison to optical assessment for polyp size measurement. This will be measured by accuracy, sensitivity, and specificity of SCALE-EYE categorization compared to optical assessment.
Sustainability | After the screening and/or surveillance colonoscopy when the endoscopist advised surveillance interval is known (on average 30 days post-colonoscopy)
  The sustainability aspect of SCALE-EYE will be assessed by exploring whether the number of colonoscopies, the colonoscopy-associated waste and carbon footprint will be reduced by correct size measurement.
Learning curve | Immediately after the screening and/or surveillance colonoscopy
  The learning curve will be evaluated by exploring the association between the number of measurements performed and the time needed for measurement and experienced difficulty.
Surveillance interval agreement | After the screening and/or surveillance colonoscopy when the endoscopist advised surveillance interval is known (on average 30 days post-colonoscopy)
  The level of agreement between the endoscopist advised surveillance interval as based on SCALE-EYE, optical assessment, and the reference standard (biopsy-forceps assisted measurement) will be compared.
(Serious) adverse events | Up to 30 days post-colonoscopy
  Serious adverse events (SAEs) and adverse events (AEs) will be summarized by proportions.

OTHER OUTCOMES:
Endoscopist experience | At baseline
  Endoscopist experience (experienced = >1000 independent colonoscopies; regular = 300 - 1000)
Age | At baseline (after informed consent is signed)
  Age in years of participant
Sex | At baseline (after informed consent is signed)
  Sex (male/female) of participant
Personal/family history of polyps or colorectal cancer (CRC) | At baseline (after informed consent is signed)
  Personal/family history of polyps or colorectal cancer (CRC) of participant - yes or no
Type of colonoscopy | At baseline (after informed consent is signed)
  Type of colonoscopy (screening or surveillance)
Type of endoscope used | During the screening and/or surveillance colonoscopy
  Type of endoscope used (SCALE-EYE equipped endoscope number)
Sedation | During the screening and/or surveillance colonoscopy
  Sedation (yes or no and which type)
Use of butyl scopolamine | During the screening and/or surveillance colonoscopy
  Use of butyl scopolamine (yes or no)
Boston Bowel Preparation Score (BBPS) | During the screening and/or surveillance colonoscopy
  BBPS (at least a score of 6 is required with a score of 2 in each colon segment)
Cecum intubation rate | At baseline
  Cecum intubation rate in percentage (%)
Polyp information | During the screening and/or surveillance colonoscopy
  Polyp location, morphology and method of polyp removal (i.e., hot/cold-snare polypectomy, EMR, ESD)
Time needed for measurement | During the screening and/or surveillance colonoscopy
  Time needed for measurement (minutes for SCALE-EYE and biopsy-forceps assisted measurement)
Experienced difficulty | During the screening and/or surveillance colonoscopy
  Experienced difficulty of SCALE-EYE measurement (scale 1-10; 1 = very easy and 10 = very difficult)
Reason of unsuccessful SCALE-EYE measurement | During the screening and/or surveillance colonoscopy
  Reasons include:
  * Unclear surroundings of polyp (i.e., feces, folds)
  * Peristalsis
  * Difficult-to-reach location
  * Mechanical difficulties (e.g. error graphic of SCALE-EYE)
  * Failed cleaning of endoscope lens/build-in laser
  * Software malfunction (freeze, crash, other)
  * Other
Withdrawal time | Immediately after the screening and/or surveillance colonoscopy
  Withdrawal time (minutes)

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - LUMC, Leiden, South Holland
  - Erasmus MC, Rotterdam, South Holland